CLINICAL TRIAL: NCT02469909
Title: Feasibility and Safety of Immediate Versus Gradual Decannulation: a Randomised Control Trial
Brief Title: Comparison Between Immediate and Gradual Decannulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaplan Medical Center (Other)
Collaborators: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Dr Oded Cohen, Dr Oded Cohen, Kaplan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENTK 34-CTIL
Record Dates: First submitted 2015-06-04; First posted 2015-06-12 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Tracheostomy
Keywords: Decannulation; tracheostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- immediate decannulation (Other): In the immediate decannulation group - the tracheostomy tube is removed and the patient would be monitored overnight in an intermediate monitored unit. On the next day a clinical evaluation would be held, and the patient would be discharge or transferred to his department according to the clinical course of the patient
  Interventions: Other: Overnight observation; Other: Pre-discharge evaluation; Other: outpatient clinic follow ups; Procedure: immediate decannulation
- Gradual tracheostomy tube decrease (Other): In the gradual decannulation group The tracheostomy tube will be reduced in 2 sizes compared with the initial inner diameter of the tube. The patients will remain with the reduced tube for 48 hours, and the tube will be removed if the patients would meet pre-decannulation evaluation
  Interventions: Other: outpatient clinic follow ups; Procedure: Gradual tracheostomy tube decrease

INTERVENTIONS:
Other: Overnight observation — patients in the immediate decannulation group would be admitted for an overnight in intensive care unit or the otolaryngology department. they would be monitored for any respiratory or airway complications.
  Arms: immediate decannulation
Other: Pre-discharge evaluation — After an overnight observation, patients in the immediate decannulation group would would undergo clinical and laboratory evaluation including vital signs and blood gases.
  Arms: immediate decannulation
Other: outpatient clinic follow ups — all patients would visit the otolaryngology outpatient clinic in 7, 30 and 90 days following decannulation for an evaluation of any respiratory complications following decannulation
Procedure: immediate decannulation — the tracheostomy tube is removed at once
  Arms: immediate decannulation
Procedure: Gradual tracheostomy tube decrease — The tracheostomy tube will be reduced in 2 sizes compared with the initial inner diameter of the tube. The patients will remain with the reduced tube for 48 hours, and the tube will be removed if the patients would meet pre-decannulation evaluation
  Arms: Gradual tracheostomy tube decrease

SUMMARY:
The investigators propose to examine the feasibility and safety of immediate (single stage) decannulation in adult patients in a controlled randomized trial. Patients who will be found fit for decannulation after an otolaryngologist and intensive care specialist assessment will be randomized into two groups: immediate decannulation and gradual decrease in cannula size. Both groups of patients will be monitored after decannulation and in the outpatient clinic for any complications following the procedure.

DETAILED DESCRIPTION:
Recruitment of the patients will be demands for decannulation evaluation of different departments in our institution. All patients who will agree to participate in the study and meet the inclusion criteria would undergo three major steps"

1. Pre decannulation evaluation by otolaryngologist and intensive care specialist following inclusion criteria.
2. Decannulation:

   In the immediate decannulation group - the tracheostomy tube is removed and the patient would be monitored overnight in an intermediate monitored unit. On the next day a clinical evaluation would be held, and the patient would be discharge or transferred to his department according to the clinical course of the patient.

   In the gradual decannulation group:

   The tracheostomy tube will be reduced in 2 sizes compared with the initial inner diameter of the tube. The patients will remain with the reduced tube for 48 hours, and the tube will be removed if the patients would meet pre-decannulation evaluation.
3. Follow up:

All patients would be followed in 7, 30, 90 days following decannulation in the outpatient clinic or in their departments if still hospitalized. In these visit questionnaires regarding possible respiratory complications will be documented.

ELIGIBILITY:
Inclusion Criteria:

Patients who underwent tracheostomy with the following conditions:

1. Tracheostomy tract is established more than 7 days
2. Normal vital signs: heart rate 50-100, 90<systolic BP <180, respiratory rate <20. Saturation >90% in room air
3. Effective cough
4. Normal swallows \ feeding possibility
5. # steps endoscopy test: through the tracheostomy tube, normal naso-laryngeal and through the tract with an upper look towards the subglottic area in order to detect subglottic stenosis.
6. Ability of the patient to breath with a capped cannula.

Exclusion Criteria:

* Patients with a major complication in tracheostomy procedure (subcutaneous emphysema, pneumothorax, bleeding, false root)
* patient with anatomical neck abnormality
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-06; Primary Completion 2018-06 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
re-insertion of the tracheostomy tube | 7 days
  number of patients who needed re-insertion of the tracheostomy tube due to respiratory distress within 7 days of decannulation
mechanical ventilation | 7 days
  number of patients who needed mechanical ventilation due to respiratory distress within 7 days of decannulation

SECONDARY OUTCOMES:
Death from any cause | 90 days
  number of patients who died from any cause within 90 days of decannulation
Respiratory distress | up to 90 fays following decannulation
  number of patients who reported difficulty breathing suggestive of stridor or by examination or intervention within 90 days of decannulation
Pneumonia | 90 days following decannulation
  number of patients who had a diagnosis of pneumonia in the period of 90 days following decannulation

CONTACTS AND LOCATIONS:
Overall Officials: Nili Segal, Dr, Principal Investigator — Soroka hospital
Locations (1):
- Kaplan medical center, Rehovot, Rehovot, Israel

REFERENCES:
- [Background] Epstein SK. Anatomy and physiology of tracheostomy. Respir Care. 2005 Apr;50(4):476-82. PMID 15807905
- [Background] Delaney A, Bagshaw SM, Nalos M. Percutaneous dilatational tracheostomy versus surgical tracheostomy in critically ill patients: a systematic review and meta-analysis. Crit Care. 2006;10(2):R55. doi: 10.1186/cc4887. PMID 16606435
- [Background] Pierson DJ. Tracheostomy and weaning. Respir Care. 2005 Apr;50(4):526-33. PMID 15807916
- [Background] Christopher KL. Tracheostomy decannulation. Respir Care. 2005 Apr;50(4):538-41. PMID 15807918
- [Background] Heffner JE. The technique of weaning from tracheostomy. Criteria for weaning; practical measures to prevent failure. J Crit Illn. 1995 Oct;10(10):729-33. PMID 10155745
- [Background] Lewarski JS. Long-term care of the patient with a tracheostomy. Respir Care. 2005 Apr;50(4):534-7. PMID 15807917
- [Result] Mitchell RB, Hussey HM, Setzen G, Jacobs IN, Nussenbaum B, Dawson C, Brown CA 3rd, Brandt C, Deakins K, Hartnick C, Merati A. Clinical consensus statement: tracheostomy care. Otolaryngol Head Neck Surg. 2013 Jan;148(1):6-20. doi: 10.1177/0194599812460376. Epub 2012 Sep 18. PMID 22990518
- [Result] De Leyn P, Bedert L, Delcroix M, Depuydt P, Lauwers G, Sokolov Y, Van Meerhaeghe A, Van Schil P; Belgian Association of Pneumology and Belgian Association of Cardiothoracic Surgery. Tracheotomy: clinical review and guidelines. Eur J Cardiothorac Surg. 2007 Sep;32(3):412-21. doi: 10.1016/j.ejcts.2007.05.018. Epub 2007 Jun 27. PMID 17588767